CLINICAL TRIAL: NCT02931149
Title: Evaluation of the Efficacy of Platelet-rich Plasma (PRP) on Advanced Endoscopic Resection Techniques
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Vicente Lorenzo-Zúñiga García, Study Principal Investigator, Germans Trias i Pujol Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EndoPRP2016
Record Dates: First submitted 2016-10-07; First posted 2016-10-12 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Platelet-rich Plasma; Endoscopic Mucosal Resection; Endoscopic Submucosal Dissection
Keywords: platelet-rich plasma; endoscopic mucosal resection; endoscopic submucosal dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Submucosal injection with PRP (Experimental): All participants in the study received submucosal injection of PRP prior to endoscopic resection
  Interventions: Drug: Platelet-rich plasma

INTERVENTIONS:
Drug: Platelet-rich plasma — Submucosal injection with PRP was performed prior to endoscopic resection
  Other Names: PRP

SUMMARY:
To avoid complications secondary to advanced endoscopic resection techniques (Endoscopic Mucosal Resection -EMR- or Endoscopic Submucosal Disection -ESD-) the endoscopists have to avoid deep thermal damage and increase mucosal healing. Platelet-rich plasma (PRP) has demonstrated efficacy in preclinical endoscopic resection models.

DETAILED DESCRIPTION:
Background:To avoid complications secondary to advanced endoscopic resection techniques (Endoscopic Mucosal Resection -EMR- or Endoscopic Submucosal Disection -ESD-) the endoscopists have to avoid deep thermal damage and increase mucosal healing. Platelet-rich plasma (PRP) has demonstrated efficacy in preclinical endoscopic resection models.

Aim: Evaluate the efficacy of PRP on participants submitted to advanced endoscopic resection techniques: EMR or ESD.

Material and Methods: The investigators have evaluated a prospective clinical study. The investigators have included 12 participants submitted to EMR or ESD. Patients were informed and accepted to participate with a written consent. Prior to endoscopy PRP was obtained from autologous blood with a comercial kit. Submucosal injection with PRP were performed prior to resection. Resection was performed with standard technique. Participants were followed-up after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic lesion higher than 40mm in diameter submitted to endoscopic resection (EMR or eSD)

Exclusion Criteria:

* Ineligibility to endoscopic resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Prevention of delayed bleeding: percentage of participants with delayed bleeding | 28 days after resection
  Delayed bleeding occurs between 13-15% of patients submitted to advanced resection techniques. The aim of this study is to evaluate the efficacy of PRP in the prevention of this complication
Prevention of coagulation syndrome (or postpolipectomy syndrome): percentage of participants with coagulation syndrome | 5 days after resection
  Coagulation syndrome occurs in around 5-7% of patients submitted to EMR or ESD. The aim is to evaluate the efficacy of PRP in the prevention of this complication

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Lorenzo-Zúñiga García, M.D., Ph.D., Principal Investigator — University Hospital Germans Trias
Locations (1):
- Endoscopy Unit. University Hospital Germans Trias, Badalona, Barcelona, Spain

REFERENCES:
- [Result] Lorenzo-Zuniga V, Boix J, Moreno de Vega V, Bon I, Marin I, Bartoli R. Efficacy of platelet-rich plasma as a shielding technique after endoscopic mucosal resection in rat and porcine models. Endosc Int Open. 2016 Aug;4(8):E859-64. doi: 10.1055/s-0042-109170. Epub 2016 Aug 10. PMID 27540573